CLINICAL TRIAL: NCT03827343
Title: Retrospective Study of Immunotherapy Related Toxicities and Factors Impacting Outcomes in Children and Adults With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919044; 19-C-N044
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-06-24

CONDITIONS: Macrophage Activation Syndrome; Primary Hemophagocytic Lymphohistiocytosis
Keywords: CAR-T Cell Therapy; Macrophage Activation Syndrome (MAS); Hemophagocytic Lymphohistiocytosis (HLH); Natural History
MeSH Terms: conditions — Macrophage Activation Syndrome; Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Retrospective chart review of children and adults with cancer enrolled on immunotherapy treatment protocols in the NCI.

SUMMARY:
Immunotherapy is changing the landscape of cancer therapy. Particularly unique to immunotherapy is the toxicity profile, which differs from chemotherapy-based strategies and can be associated with inflammatory responses and/or autoimmune type reactions resulting from activation of the immune system. Referred to as immune related adverse events (irAEs), these adverse events may require systemic immunosuppression or have other consequences and present unique management challenges. Specific to CAR T-cell and other adoptive cell therapies is the constellation of symptoms referred to as cytokine release syndrome (CRS), which can range in severity from mild to severe, and can require both cytokine directed blockade and/or systemic immunosuppression to ameliorate the side effects. While side effects may be unique to each individual immunotherapy, and may also be patient specific, cumulative experience will help to inform toxicity profiles and improve management of side effects and overall outcomes.

Given the number of immunotherapeutic approaches at the NCI, the primary goal of this protocol is to facilitate retrospective chart review of various immunotherapy trials at the NCI used in the treatment of cancer to comprehensively study toxicity profiles. This study will not involve the use of specimens or participant contact. All data that is needed has already been collected on the individual treatment protocols and is available in CRIS records or protocol specific databases.

Data will only be collected from treatment protocols where the PI has given permission for use of the data on the trial the subject was enrolled on. This protocol will be amended to incorporate new research objectives and new protocols as necessary.

DETAILED DESCRIPTION:
Immunotherapy is changing the landscape of cancer therapy. Particularly unique to immunotherapy is the toxicity profile, which differs from chemotherapy-based strategies and can be associated with inflammatory responses and/or autoimmune type reactions resulting from activation of the immune system. Referred to as immune related adverse events (irAEs), these adverse events may require systemic immunosuppression or have other consequences and present unique management challenges. Specific to CAR T-cell and other adoptive cell therapies is the constellation of symptoms referred to as cytokine release syndrome (CRS), which can range in severity from mild to severe, and can require both cytokine directed blockade and/or systemic immunosuppression to ameliorate the side effects. While side effects may be unique to each individual immunotherapy, and may also be patient specific, cumulative experience will help to inform toxicity profiles and improve management of side effects and overall outcomes.

Given the number of immunotherapeutic approaches at the NCI, the primary goal of this protocol is to facilitate retrospective chart review of various immunotherapy trials at the NCI used in the treatment of cancer to comprehensively study toxicity profiles. This study will not involve the use of specimens or participant contact. All data that is needed has already been collected on the individual treatment protocols and is available in CRIS records or protocol specific databases. Data will only be collected from treatment protocols where the PI has given permission for use of the data on the trial the subject was enrolled on or from standard of care protocols. This protocol will be amended to incorporate new research objectives and new protocols as necessary.

ELIGIBILITY:
* Retrospective chart review of various immunotherapy trials at the NCI used in the treatment of cancer to comprehensively study toxicity profiles. This study will not involve the use of specimens or participant contact. All data that is needed has already been collected on the individual treatment protocols and is available in CRIS records or protocol specific databases.

Ages: 1 Month to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with cancer enrolled on immunotherapy treatment protocols in the NCI.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To develop a retrospective study to allow for comparison of immunotherapy related toxicity profiles and risk factors across a set of protocols in the NCI. | 2 years
  Summary of immunotherapy related toxicity profiles and risk factors across a set of protocols in the NCI.

SECONDARY OUTCOMES:
Evaluate infectious complications and their risk factors in patients who receive CAR-T cell therapy for cancer | 2 years
  Summary of infectious complications and their risk factors in patients who receive CAR-T cell therapy for cancer
Evaluate the incidence, risk factors for, and treatment of HLH/MAS (now renamed IEC-HS) in patients who receive CAR-T cell therapy. | 2 years
  Incidence and treatment of HLH/MAS (now renamed IEC-HS) in patients who receive CAR-T cell therapy
Incidence and time to resolution | 2 years
  Incidence of and time to resolution of grade 3 and 4 cytopenias post-CAR T-cell therapy in those who achieve a complete remission.
Overall and relapse free survival | 2 years
  Summary of overall and relapse free survival and transplant associated toxicities for patients undergoing HSCT following CAR-T cell therapy
Incidence of end organ toxicities | 2 years
  Incidence of grade 3 and 4 end organ toxicities experienced within the first 30 days of CAR T-cell therapy and includes associations between pre-CAR organ function as well as post-CAR response to such toxicities as well as validate the CAR-Comorbidity Index as predictive model of CRS severity
Evaluate response and toxicity profile of second CAR T-cell infusions | 2 years
  Summary of factors associated with response to second CAR T-cell infusion
Evaluate impact of race/ethnicity and obesity on CAR T-cell outcomes | 2 years
  Summary of response and toxicity profiles in patients based on race/ethnicity and also in those who are obese compared to those who are not.
Evaluate impact of cryopreservation on outcomes following CAR T-cell infusion | 2 years
  Summary of cryopreservation and patients' outcomes following CAR T-cell infusion
Evaluate outcomes for patients with ALL and Down Syndrome following CAR T-cell therapy | 2 years
  Summary of outcomes of patients with ALL and Down Syndrome who have received CAR T-cell therapy
Evaluate absolute lymphocyte count following lymphodepleting chemotherapy | 2 years
  Summary of absolute lymphocyte count across lymphodepleting regimens
Evaluate relationship between clinical variable and apheresis and manufacturing products | 2 years
  Summary of clinical variables and apheresis and manufacturing products
Evaluate incidence of hypertension, identify risk factors for development of hypertension, summarize medical management in CAR setting, and identify complications | 2 years
  Summary of incidence of hypertension, risk factors, medical management and complications
Describe baseline demographics, prior treatment characteristics and outcomes based on patients who are referred to CAR T-cell program | 2 years
  Summary of demographics, prior treatment and outcomes for patients referred to CAR T-cell program
Incidence of pre-infusion BCA and use of BCA as a prognostic marker for CAR T-cell associated toxicity and efficacy | 2 years
  Incidence of BCA pre-infusion and use as a prognostic marker for CAR T-cell associated toxicity and efficacy
Presence and durability of CD72 expression in both B-ALL and normal B-ALL/hematogones | 2 years
  Summary of CD72 expression in both B-ALL and normal B-ALL/hematogones and evaluate use as prognostic marker for CAR T-cell associated toxicity and efficacy
Evaluate interventions, documentation of care goals, and use of palliative care consultation or other symptom management | 2 years
  Summary of interventions, documentation of care goals, and use of palliative care consultation or other symptom management for patients treated with CAR T-cell therapy
Evaluate long-term outcomes of survivors who received CAR T-cell therapy | 2 years
  Summary of long-term outcomes of survivors who received CAR T-cell therapy
Evaluate cross compare responses and outcomes based on NGS MRD and FC MRD | 2 Years
  Summary of cross compare responses and outcomes based on NGS MRD and FC MRD
Evaluate the role of manufacturing changes on CAR T-cell outcomes | 2 Years
  Summary of the role of manufacturing changes on CAR T-cell outcomes
Evaluate the impact of clonal hematopoiesis on CAR T-cell outcomes | 2 Years
  Summary of the impact of clonal hematopoiesis on CAR T-cell outcomes
Evaluate CAR T-cell related coagulopathies | 2 Years
  Summary of CAR T-cell related coagulopathies
Evaluate the use of anti-cytokine therapy to treat toxicities after CAR T-cell infusion | 2 Years
  Summary of the use of anti-cytokine therapy to treat toxicities after CAR T-cell infusion
Evaluate outcomes of CAR T-cells in patients with extramedullary disease | 2 Years
  Summary of outcomes of CAR T-cells in patients with extramedullary disease

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Derived] Culbert AA, Gava F, Valtis YK, Satta T, Vora S, Rocco JM, Nussenblatt V, Silbert SK, Shalabi H, Yates B, Park JH, Lamble AJ, Rejeski K, Shah NN. Pre-infusion risk factors predict severe infectious complications of CAR T-cell therapy in pediatric and adult patients with B-ALL. J Immunother Cancer. 2025 Sep 14;13(9):e012436. doi: 10.1136/jitc-2025-012436. PMID 40953923
- [Derived] Silbert SK, Madan S, Holland EM, Steinberg SM, Little L, Foley T, Epstein M, Sarkisian A, Lee DW, Nikitina E, Kakumanu S, Ruppin E, Shalabi H, Yates B, Shah NN. A comprehensive analysis of adverse events in the first 30 days of phase 1 pediatric CAR T-cell trials. Blood Adv. 2023 Sep 26;7(18):5566-5578. doi: 10.1182/bloodadvances.2023009789. PMID 37486616
- [Derived] Holland EM, Yates B, Steinberg SM, Yuan CM, Wang HW, Annesley C, Shalabi H, Stroncek D, Fry TJ, Krueger J, Jacoby E, Hsieh E, Bhojwani D, Gardner RA, Maude SL, Shah NN. Chimeric Antigen Receptor T Cells as Salvage Therapy for Post-Chimeric Antigen Receptor T Cell Failure. Transplant Cell Ther. 2023 Sep;29(9):574.e1-574.e10. doi: 10.1016/j.jtct.2023.06.019. Epub 2023 Jun 30. PMID 37394115